CLINICAL TRIAL: NCT04996498
Title: Hemostatic Effect of Intrauterine Instillation of Oxytocin in Hysteroscopic Myomectomy: A Randomized Double Blinded Control Trial
Brief Title: Hemostatic Effect of Intrauterine Instillation of Oxytocin in Hysteroscopic Myomectomy
Acronym: oxytocin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amir Hamdy Abd El hady Mahfouz, assistent lecturer, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Hysteroscopic Myomectomy:
Record Dates: First submitted 2021-07-07; First posted 2021-08-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Leiomyoma
Keywords: Hysteroscopic Myomectomy
MeSH Terms: conditions — Leiomyoma | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized controlled double blinded clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The allocation will be concealed in sealed, sequentially numbered, white envelopes which will be prepared by a statistician where the drug will be covered with adhesive tape and handed over to the data collector. each woman will collect the corresponding sealed envelope directly from the data collector and it will be opened just before application of the drug.
  the surgeon, the assistant and the nurse performing the procedure and the patient will be blinded to the medication drug which will be used inside the distention medium.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Oxytocin group): (Active Comparator): 30 women will undergo a hysteroscopic myomectomy with the use of 10 IU of oxytocin for every 1000 ml of the distending medium (1,5% Glycine ).
  Interventions: Drug: Oxytocin
- Group B (Placebo group): (Placebo Comparator): 30 women will undergo hysteroscopic myomectomy with the use of a sterile bacteriostatic water ampule in the distending medium (1,5% glycine).
  Interventions: Other: sterile bacteriostatic water ampule

INTERVENTIONS:
Drug: Oxytocin — intrauterine Instillation of oxytocin in distention media used during Hysteroscopic Myomectomy
  Other Names: syntocinon
  Arms: Group A (Oxytocin group):
Other: sterile bacteriostatic water ampule — a placebo drug similar in shape to oxytocin ampules
  Arms: Group B (Placebo group):

SUMMARY:
There is no previous study on the hemostatic effect of intrauterine instillation of oxytocin in hysteroscopic myomectomy. All previous studies focused on intravenous administration of oxytocin.

This trial may modify the surgical environment in hysteroscopic myomectomy by decreasing intraoperative bleeding to a degree that the amount of distention medium required for uterine distention will be reduced with a better visibility and shorter operation time.

The standard treatment of symptomatic myomas is hysterectomy for women who have completed childbearing period, and myomectomy for women who wish to preserve fertility hysteroscopic myomectomy currently is the gold standard minimally invasive procedure for the management of symptomatic submucous fibroids. Success of hysteroscopic myomectomy depends on good visualization throughout the procedure, via the correct distending pressure, continuous irrigation and the use of electrosurgery to control bleeding. Prolonged procedures that need continuous irrigation under high pressure are associated with higher risk of excessive fluid absorption and intravasation syndrome due to opened blood vessels within the myometrial, moreover, the thermal damage of the healthy tissues is increased with the use of the coagulation current.

Oxytocin receptors exist in the non-pregnant uterus but the concentration of the receptors is much lower than in pregnancy. this is why the clinical use of oxytocin outside of pregnancy is limited Oxytocin acts on oxytocin receptors in the myometrium and fibroid tissue leading to uterine contraction and constriction of uterine vasculature due to uterine contraction and vaso-constrictive effect of oxytocin thus reducing uterine perfusion and results in reducing intraoperative bleeding.

DETAILED DESCRIPTION:
Patients will be subjected to:

1. History taking: including personal history, menstrual and obstetric history, medical and surgical history, medications.
2. Clinical examination; General and local with special concern about:

   1. Size and position of the uterus
   2. Transvaginal ultrasound to determine the number, size, location of fibroids and evaluation of the myometrial free margin that is defined as the minimum thickness between the outer edge of the fibroid and the inner edge of uterine serosa.
3. Laboratory evaluation: All participants will have routine blood tests: Complete Blood Count (CBC), serum creatinine, viral markers, coagulation profile and liver function tests.

Surgical procedure:

1. Office hysteroscopy will be performed the day before the procedure with the use of a 2-9 mm telescope with continuous-flow sheath (Hopkins II telescope 30 degrees: Karl storz) to assess and confirm the fibroid location, its intracavitary portion and to exclude any associated uterine pathology).
2. Hysteroscopy will be performed in the early proliferative phase (postmenstrual) in dorsal lithotomy position under general anesthesia, cervical dilatation will be done with Hegar dilators then resection of the submucous fibroid using monopolar resectoscope using 1,5% glycine as a distension medium by single operator to avoid inter-observer variability.
3. The intervention group (oxytocin group) will receive 10 IU of oxytocin for every 1000 ml of the distending medium (1,5% Glycine). While in the control group a sterile bacteriostatic water ampule in the same form will be added to every 1000 ml of the distending medium (1,5% Glycine).
4. After completing the procedure, the surgeon will complete a record scale to document estimated blood loss, rating the bleeding (0: no bleeding, I; mild bleeding, II: moderate bleeding, III: severe bleeding, IV: severe bleeding with clots). Also will document the clarity of visual field using 3 point likert scale as (poor, fair, good).
5. Post operative settings:

   * the duration of surgery and the volume of injected media will be calculated and documented.
   * all patients will be subjected to postoperative hemoglobin 24 hours after the procedure, any intraoperative or postoperative complications will be documented

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic patient (Menorrhagia, recurrent pregnancy loss or infertility).
2. 1 or 2 submucous uterine myoma diagnosed by ultrasound with a diameter less than 4 cm
3. Myoma with FIGO 0 or 1.
4. Body mass index less than 35.

Exclusion Criteria:

1. Pregnancy
2. Active pelvic infection
3. history of bleeding disorder or patient on anti-coagulant.
4. hepatic and renal diseases.
5. history of ischemic heart disease.
6. Patients with uterine structural abnormality or uterine septum.
7. Present or history of cervical or uterine cancer.
8. Preoperative administration of gonadotropin-releasing hormone analogues or danazol.
9. Allergy to glycine.
10. Patients with hypercoagulopathy.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
the change in hemoglobin level 24 hours after the procedure surgery | preoperative and 24 hour postoperative
  the change of hemoglobin postoperative to know the effect of oxytocin compared to placebo in reducing blood loss.
  surgery compared to the pre-operative values to see if intrauterine instillation of oxytocin will reduce blood loss during hysteroscopic myomectomy
the change of hematocrit level 24 hour after the procedure | preoperative and 24 hour postoperative
  a follow up CBC is done 24 hour after the procedure to see the difference in hematocrit and know about the blood loss intraoperative

SECONDARY OUTCOMES:
the surgeon rating of intraoperative bleeding and the visual field quality of operative view, | immediately postoperative
  After completing the procedure, the surgeon will complete a record scale to document estimated blood loss, rating the bleeding (0: no bleeding, I; mild bleeding, II: moderate bleeding, III: severe bleeding, IV: severe bleeding with clots).
the duration of surgery, intraoperative | immediately postoperative
  Success of hysteroscopic myomectomy depends on good visualization throughout the procedure, so, if oxytocin decrease blood loss intraoperative , the operation time will be reduced .
intraoperative and postoperative complications | intraoperative and within the first 24 hours postoperative
  there are some operative complications as uterine perforation , cervical tear and fluid overload also, there is some adverse effects of oxytocin as arrythmia, nausea, vomiting , hypotension and abdominal pain
the surgeon rating the visual field | immediately postoperative
  After completing the procedure, the surgeon will document the clarity of visual field using 3 point scale as (poor, fair, good)
the volume of distension media used intraoperative | immediately postoperative
  glycine 1,5% is used as a distention media during procedure, each solution contain 1000 ml . counting the number of solution used intraoperative to calculate the amount of distension media used.

CONTACTS AND LOCATIONS:
Overall Officials: amir Mahfouz, Master, Principal Investigator — AinShams MH
Locations (1):
- Ain shams university maternity hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Spiezio Sardo A, Mazzon I, Bramante S, Bettocchi S, Bifulco G, Guida M, Nappi C. Hysteroscopic myomectomy: a comprehensive review of surgical techniques. Hum Reprod Update. 2008 Mar-Apr;14(2):101-19. doi: 10.1093/humupd/dmm041. Epub 2007 Dec 6. PMID 18063608
- [Background] Vilos GA, Allaire C, Laberge PY, Leyland N; SPECIAL CONTRIBUTORS. The management of uterine leiomyomas. J Obstet Gynaecol Can. 2015 Feb;37(2):157-178. doi: 10.1016/S1701-2163(15)30338-8. PMID 25767949
- [Background] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435
- [Background] Maggi M, Magini A, Fiscella A, Giannini S, Fantoni G, Toffoletti F, Massi G, Serio M. Sex steroid modulation of neurohypophysial hormone receptors in human nonpregnant myometrium. J Clin Endocrinol Metab. 1992 Feb;74(2):385-92. doi: 10.1210/jcem.74.2.1309835.
- [Background] Atashkhoei S, Fakhari S, Pourfathi H, Bilehjani E, Garabaghi PM, Asiaei A. Effect of oxytocin infusion on reducing the blood loss during abdominal myomectomy: a double-blind randomised controlled trial. BJOG. 2017 Jan;124(2):292-298. doi: 10.1111/1471-0528.14416. Epub 2016 Nov 15. PMID 27862855
- See also: practice guidelines for the diagnosis and management of submucous leiomyomas. Journal of minimally invasive gynecology, — https://doi.org/10.1016/j.jmig.2011.09.005